CLINICAL TRIAL: NCT03647592
Title: Real World Study to Evaluate the Efficacy and Resistant Mechanism of Erlotinib/Gefitinib Combined With Bevacizumab in First Line EGFR Mutation Positive Advanced Non-aquamous Non-small Cell Lung Cancer
Brief Title: Real World Study on Erlotinib/Gefitinib Combined With Bevacizumab in Advanced Non-aquamous Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, professor, Hunan Province Tumor Hospital
Other Study IDs: WECAN
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Bevacizumab; Erlotinib/Gefitinib; EGFR mutation positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohorts 1: patients with EGFR mutation-positive who received treatment of Erlotinib/Gefitinib Combined With Bevacizumab
  Interventions: Drug: Erlotinib/Gefitinib combined with Bevacizumab

INTERVENTIONS:
Drug: Erlotinib/Gefitinib combined with Bevacizumab — Erlotlnib,150mg po qd/gefitinib 250mg po qd +Bevacizumab(15mg/kg),lvgtt,every 21 day ,evaluate every 2 months
  Other Names: treatment of A+T

SUMMARY:
This study aims to explore the efficacy and safety of Erlotinib/Gefitinib combined with bevacizumab in the real world for advanced non-squamous cell lung cancer with EGFR mutation, explore new drug resistance mechanisms under the A+T regimen and consistency between plasma and tissue detection driving genes, and finally assess the predictive value of plasma dynamic detection driving gene mutation profiles in predicting disease. The role of disease progression risk.

DETAILED DESCRIPTION:
A retrospective study of 30 cases of advanced non-squamous non-small cell lung cancer (NSCLC) with EGFR mutation positive treated with A+T was conducted to observe the efficacy and safety of A+T regimen in the real world. Exploratory research contents are as follows: 1. Consistency between tissue gene test (NGS) and plasma gene test (NGS) at the initial diagnosis; 2. Consistency between tissue gene test (NGS) and plasma gene test (NGS) at the progression of A + T treatment; 3. New drug resistance mechanism of A + T treatment; 4. Plasma dynamics during A + T treatment. Detection (the first efficacy evaluation and a blood sampling before imaging PD) exploration and imaging progress sequence; 5. Plasma large panel dynamic drive gene mutation spectrum analysis to build disease progression risk model.

ELIGIBILITY:
Inclusion Criteria:

* EGFR mutation(19del/L858R)
* advanced non-saquamous non-small cell lung cancer
* primary treatment of first diagnosis
* performance status（0-1)

Exclusion Criteria:

* other genes mutation
* saquamous

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 non-saquamous non-small cell lung cancer with EGFR mutation positive (19del/L858R) were inrolled in this study.
  ECOG PS 0-1 All the patients recieved the treatment of erlotinib combined with Bevacizumab.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Approximately 1 years
  Progression free survival

SECONDARY OUTCOMES:
OS | Approximately 1 years
  Overall survival
DCR | Approximately 1 years
  Disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincal Tumor Hospital, Changsha, Hunan, China